CLINICAL TRIAL: NCT02053207
Title: The Cog-Train Feasibility Study: a Single-arm Trial Investigating the Feasibility of a Preoperative Cognitive Training Intervention (Cog-Train) in Cardiac Surgical Patients
Brief Title: Feasibility Study of Preoperative Cognitive Training in Cardiac Surgical Patients
Acronym: Cog-Train
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Medical Research Council Cognition and Brain Sciences Unit (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P01907
Record Dates: First submitted 2014-01-20; First posted 2014-02-03 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: Cognitive training; Brain training; Plasticity-based training; Cardiac surgery; Preoperative; Cognitive function
MeSH Terms: conditions — Postoperative Cognitive Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cog-Train Intervention (Experimental)
  Interventions: Behavioral: Cog-Train Intervention

INTERVENTIONS:
Behavioral: Cog-Train Intervention — Twenty-one days prior to surgery, patients will begin self-administering the intervention using an iPad tablet. This intervention will consist with daily sessions of at least 20 minutes of the Cog-Train task (the task and regimen used to obtain robust effects in previous studies by members of our group). Cog-Train is an n-back task - an adaptive working memory computer game that extends players' working memory capacity by getting progressively more difficult as the player's performance increases.

SUMMARY:
The purpose of this study is to evaluate the feasibility of administering a 20-day preoperative cognitive training intervention (Cog-Train) to a widely inclusive sample of cardiac surgical patients.

DETAILED DESCRIPTION:
Cognitive outcomes remain poor after cardiac surgery. Data from the field of cognitive neuroscience suggests that cognitive training, which harnesses the brain's adaptive plasticity to improve, maintain, or restore function in a target area, can be used to strengthen brain resilience and improve cognitive outcomes following challenge. While its effectiveness has been demonstrated in older adults as well as in other (nonsurgical) patient populations, no training intervention like this has ever before been used in any surgical patient in the preoperative period. The purpose of this study is to evaluate the feasibility of administering a 20-day cognitive training intervention (Cog-Train) to a widely inclusive sample of cardiac surgical patients before their surgery. Data obtained will be used to design a full-scale randomised controlled trial (RCT) on Cog-Train's effectiveness in improving postoperative cognitive outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective cardiac surgery with cardiopulmonary bypass at Papworth Hospital
* Aged 60+ years

Exclusion Criteria:

* Surgery scheduled for sooner than 21 days
* 'Off-pump' surgery being considered
* Inability to obtain informed consent
* Sensory or motor impairments impeding use of task
* Communication barriers impeding administration of study procedures
* Inability to demonstrate understanding of task and/or study procedures
* Inability to make time commitment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Training performance gain | From 21 days prior to scheduled surgery to 1 day prior to scheduled surgery
  Average increase in training task level achieved from first to last training day
Adherence to training regimen | From 21 days prior to scheduled surgery to 1 day prior to scheduled surgery
  Mean number of training days completed according to instructions

SECONDARY OUTCOMES:
Recruitment and retention | 10 weeks
  Proportion of patients approached who can do the task and are willing to take part
Satisfaction and acceptability | At 1 day prior to scheduled surgery
  Self report questionnaire
Side-effects | From 21 days prior to scheduled surgery to up to 14 days after surgery
  Side effects and severity reported by patients and proportion of patients who reported side-effects

CONTACTS AND LOCATIONS:
Overall Officials: Alain Vuylsteke, MD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schweizer S, Hampshire A, Dalgleish T. Extending brain-training to the affective domain: increasing cognitive and affective executive control through emotional working memory training. PLoS One. 2011;6(9):e24372. doi: 10.1371/journal.pone.0024372. Epub 2011 Sep 19. PMID 21949712